CLINICAL TRIAL: NCT00271232
Title: InSync III Marquis Model 7279 Cardioverter Defibrillator Cardiac Resynchronization System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 199
Record Dates: First submitted 2005-12-28; First posted 2005-12-30 (Estimated); Last update posted 2007-12-21 (Estimated); Status verified 2007-12

CONDITIONS: Heart Failure
Keywords: Heart Failure, Cardiac Resynchronization
MeSH Terms: conditions — Heart Failure | interventions — Cardiac Resynchronization Therapy

INTERVENTIONS:
Device: Cardiac resynchronization therapy

SUMMARY:
People who have a dangerously fast heart beat, or whose heart is at risk of stopping beating, may be in need of an electronic device called an implantable cardioverter defibrillator (ICD). An ICD is implanted surgically just under the skin in the upper chest area and it sends a strong electrical impulse, or shock, to the heart to return it to a normal rhythm. If the heart is beating too slowly or at an abnormal rhythm, an ICD can also pace the heart to return the heart to its normal rhythm.

The InSync III Marquis device can change the timing of when the left and right ventricles of the heart are paced to beat. This is called "V to V timing". V to V timing may further improve the pumping function of the heart. The purpose of this study is to determine whether or not this V to V timing feature of the InSync III Marquis system is safe and effective.

ELIGIBILITY:
Inclusion Criteria:

Subject has, or is at risk of having, a heart beat that is too fast and his/her doctor has determined the need for an implantable cardioverter defibrillator.

Subject is on optimal medical treatment for heart failure.

Subject has reduced left ventricular ejection fraction (LVEF≤35%). (LVEF is a measurement of how well the left ventricle pumps blood out to the rest of the body. The higher the LVEF the more blood the ventricle is pumping.)

Subject who has heart failure which severely limits daily activities (NYHA Class III) or subject who has severe heart failure and should always be resting (NYHA Class IV)

Subject who has a QRS≥130ms (The QRS interval is a measurement of how the electrical signal involved in a heart beat travels/conducts through the ventricles. A wide QRS (more than 120 ms) suggests that there is a conduction problem (or block) in the ventricles.)

Subjects with a left ventricular end diastolic dimension (LVEDD≥55mm). (The LVEDD is a measurement taken during an echocardiogram that is one indication of the health of the left ventricle.)

Exclusion Criteria:

Subject has unstable chest pain, heart surgery within past 3 months

Subject has liver function tests greater than 3 times normal limits

Subject has chronic (permanent) atrial arrhythmias (fast heart beats in the upper chamber(s) of the heart)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238
Dates: Start 2003-03; Study Completion 2005-04

PRIMARY OUTCOMES:
To evaluate the safety and effectiveness of the InSync III Marquis Model 7279 in heart failure patients who were indicated for an ICD

SECONDARY OUTCOMES:
Rate of oxygen uptake (consumption) measured during exercise, all adverse events, echocardiographic assessments (tests done using ultra sound to examine the health of the heart), and device performance

CONTACTS AND LOCATIONS:
Locations (34):
- United States (34):
  - Anchorage, Alaska
  - Phoenix, Arizona
  - Los Angeles, California
  - Stanford, California
  - Jacksonville, Florida
  - Pensacola, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Beech Grove, Indiana
  - Burlington, Massachusetts
  - Minneapolis, Minnesota
  - Saint Paul, Minnesota
  - Kansas City, Missouri
  - Lincoln, Nebraska
  - Las Vegas, Nevada
  - Lebanon, New Hampshire
  - New York, New York
  - Rochester, New York
  - Syracuse, New York
  - Raleigh, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Lancaster, Pennsylvania
  - Philadelphia, Pennsylvania
  - Wynnewood, Pennsylvania
  - Aiken, South Carolina
  - Columbia, South Carolina
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Falls Church, Virginia
  - Milwaukee, Wisconsin

REFERENCES:
- [Derived] Abraham WT, Leon AR, St John Sutton MG, Keteyian SJ, Fieberg AM, Chinchoy E, Haas G. Randomized controlled trial comparing simultaneous versus optimized sequential interventricular stimulation during cardiac resynchronization therapy. Am Heart J. 2012 Nov;164(5):735-41. doi: 10.1016/j.ahj.2012.07.026. Epub 2012 Oct 2. PMID 23137504